CLINICAL TRIAL: NCT04165655
Title: Keep Achieving:The Impact of Group Based Activity Programmes on Children Who Have Autism and Their Families
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Midlands Psychology CIC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MP/KA-1
Record Dates: First submitted 2019-11-08; First posted 2019-11-18 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum condition; ASC; Children and young people; Social skills; Problem behaviours; Activity intervention; Wellbeing; Self image; Social connectedness
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills

STUDY DESIGN:
Intervention Model Description: The study will use a between-subject design where by participants will be assigned to either the experimental (10-week programme) or waitlist control group. Participants will be assigned a group based in the area in which they live. As the 10-week programme will be running in Tamworth, those participants living in Tamworth and surrounds will be assigned to the experimental group. The participants living in Cannock and surrounds will be assigned to the waitlist control group and participate in a 10-week programme after this research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Keep Achieving (KA) group (Experimental): Participants in the experimental group will take part in a 10-week group based activity programme. The activity programme will consist of 1, 50 minute session each week for the duration of 10-weeks. The activity sessions will include semi-structures free play sessions, sport specific sessions facilitated by local sports teams and swimming sessions.
  Interventions: Behavioral: Keep Achieving (KA)
- Waitlist control group (No Intervention): Participants in this group will not receive the 10-week group based activity intervention throughout the duration of this study. Participants will be able to participate in the 10-week activity intervention once this research has ended.

INTERVENTIONS:
Behavioral: Keep Achieving (KA) — The 10-week group based activity programme will consist of 10 sessions each lasting 50 minutes.
  Other Names: 10-week group based activity programme
  Arms: Keep Achieving (KA) group

SUMMARY:
Participation in structured activities and physical activity (PA) have been linked to several indicators of positive development such as self-esteem and psychological health as well as greater academic outcomes and lower school drop-out rates. Despite this, 77% of boys and 80% of girls aged 5-15 in the UK also fall below the national physical activity guidelines of 60 minutes of moderate to vigorous activity per day.

Children with Autism Spectrum Conditions (ASC) may be at particular risk for inactivity as they are more likely to experience barriers to participation in these types of activities and motor skills impairments, common in people with ASC, can further limit participation in PA. Studies that have attempted to increase PA in young people with autism have shown reduction in problem behaviours such as inattention and aggression and increase in positive behaviours such as sleep, improvements in quality of life, academic performance and physical competence, and reductions in stress.

The primary research aim is to investigate whether participation in a 10-week group based activity programme affects social skills and problem behaviours in CYP with ASC. It is hypothesised that children and young people (CYP) participating in the 10-week group based activity programme will show greater improvements in social skills and a greater reduction in problem behaviours than CYP not participating in the 10-week activity programme (control condition).

Participants will be assigned to either the experimental condition (10-week activity programme) or waitlist control group. Participants in the 10-week activity programme will participate in group based activities including; 'pick up and play' sessions, swimming sessions and sport specific sessions coached by local sports teams. The 10-week activity programme consists of 1, 50 minute session per week for 10-weeks.

Questionnaire data will be collected pre and post intervention to see if there are any differences in social skills and problem behaviour scores between the experimental and control group for CYP with ASC.

DETAILED DESCRIPTION:
Background:

Participation in structured activities and physical activity (PA) have been linked to several indicators of positive development such as self-esteem and psychological health as well as greater academic outcomes and lower school drop-out rates. Despite this, 77% of boys and 80% of girls aged 5-15 in the UK also fall below the national physical activity guidelines of 60 minutes of moderate to vigorous activity per day.

Children with Autism Spectrum Conditions (ASC) may be at particular risk for inactivity as they are more likely to experience barriers to participation in these types of activities and motor skills impairments, common in people with ASC, can further limit participation and enjoyment in PA and structured activities such as sports clubs and swimming lessons. Studies have shown that even at a young age children with ASC are less active than non-ASC children, and this physical activity gap gets wider as children get older.

Studies that have attempted to increase PA in young people with autism have shown reduction in problem behaviours such as inattention and aggression and increase in positive behaviours such as sleep, improvements in quality of life, academic performance and physical competence, and reductions in stress. However, many of these studies only worked with children 1:1 and therefore little is known about group-based activity intervention in young people with ASCs which could provide people with ASC opportunities to be physically active and as well as opportunities to socialise with others.

Parental modelling has been shown to be a predictor of children's PA behaviours with a positive correlation between adult and child PA levels. Given the influential role parents play on children's PA behaviours, parental involvement could be used as a function to increase PA in children with ASC.

It is not only young people with ASC who may struggle to access or fail to participate in sufficient PA but adults of the so called 'normal population'. In the UK, 34% of men and 42% of women do not meet the UK physical activity guidelines of 150 minutes of moderate activity per week. PA and civic participation may be particularly beneficial to parents of children with ASC as parents of children with developmental disorders have been shown to report lower quality of life, more depression, and greater pessimism about the future than parents of typically developing children. Caring for a child with a developmental disorder can also be more time consuming and costly. As a result this parents with children who have ASC may experience lower sense of connectedness to the social world and may experience loneliness, anxiety and low self-esteem.

Aims:

To investigate whether participation in a 10-week group based activity programme affects social skills and problem behaviours in CYP with ASC

Secondary aims:

To investigate the effects of a weekly group based activity programme on parental wellbeing and social connectedness.

To investigate parental goals for participating in a group based activity programme and evaluate progress toward these goals at the end of the programme.

To investigate the effects of a weekly group based activity programme on the self image of children with an ASC.

Hypotheses:

There will be a greater improvement in social skills and a reduction in problem behaviours in CYP participating in the group based activity programme than those in the waitlist control group.

An increase in parental wellbeing and social connectedness in parents participating in the group based activity programme than those parents in the waitlist control group.

Method;

Participants:

The sample will consist of 40 CYP with an ASC and 40 parents/carers of CYP with an ASC. 20 CYP with ASC and 20 parents/carers will be assigned to the experimental condition, participating in the 10-week group based activity programme, and 20 CYP with ASC and 20 parents/carers will be assigned to the waitlist control group. Principle inclusion criteria include; children with a working or full ASC diagnosis aged between 8 -12 years, self-declared physical wellbeing to participate in activities. Siblings and additional adults will also be invited to participate in the programme in order to support their sibling with ASC and to make attendance easier for parents who would otherwise struggle with childcare if they were not able to participate in the programme as a family. However, data will not be collected from this group. Participants will be recruited through advertisements on social media and at local autism support groups.

Design:

The study will use a between subjects design. Participants will be allocated to either the experimental group, 10-week group based activity programme, or the waitlist control group. The 10-week group based activity programme will consist of 10 sessions each lasting 50 minutes.

4 of these sessions will be semi-structured free play sessions with a range of activities taking place in order to refresh and sustain interest each week. Specific activities will be selected for sessions that are associated with key areas of difficulty related to the autistic triad of impairments. This means that behind each activity here will be a main focus to encourage either social interaction, provide sensory feedback, or target specific motor skills. These activities will include soft archery, hockey, football, obstacle courses, trampolining, volleyball, frisbee, glow in the dark activities and crafts.

3 events will be facilitated by sports clubs i.e handball, football, rugby and will be similarly divided up into different activities on the day to sustain interest. For instance, football would be broken down into passing skills, dribbling, shooting, and a small game.

2 sessions take place in the swimming pool and families will have access to floats and inflatable balls.

1 session will be a novel activity such as a climbing session at a 'clip and climb' to celebrate participation in the programme.

Procedure:

Participants will be recruited via online advertisements. These advertisements will target families living within the Tamworth and Cannock vicinity. The advertisements will inform prospective participants of the 10-week group based programme and ask all interested to contact the research team for further information. All interested participants will be informed that a 10-week programme is due to run in Tamworth from approximately January - March and in Cannock from April - June.

Participants will be sent (via email) an information sheet detailing what the study entails and the consent forms to be completed for all those taking part in the research. Participants will be informed that they can drop out of the study at anytime and ask for their data to be withdrawn. Participants will also have the opportunity to contact the researchers and have any queries addressed.

Once consent has been obtained from all participants, they will be assigned to either the experimental group (participating in the 10-week activity programme) or the waitlist control group. Participants will be assigned a group based on their location. Participants living within the Tamworth area will be assigned to the experimental group as this is the location in which the first 10-week programme is taking place. Participants living within the Cannock area will be assigned to the waitlist control group and take part in the 10-week programme at a later date. 3 weeks prior to the start of the activity programme, all participants will be sent the Social Skills Improvement System (SSIS), Social Connectedness Scale - Revised (SCS-R), Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS), the Self Image Profile (SIP) and goal based outcomes (GBO) measure and asked to return all of these prior to the start of the 10-week activity programme. Once the 10-week activity programme has ended, participants in both the experimental and control groups will again be asked to complete the SSIS, SCS-R, SWEMWBS, SIP and GBOs. Participants will be thanked for their participation in the study and those in the waitlist control group will be enrolled onto the next 10-week activity programme.

Results;

Proposed data analysis:

A one-way MANOVA will be used to compare the scores for social skills and problem behaviours on the parental SSIS and child SSIS.

Scores from the SCS-R and SWEMWBS will also be compared between the experiment and control group using a one-way MANOVA.

The GBO ratings from pre and post intervention for the experimental group will be compared to investigate to what extent parents felt their goals for participation were reached.

Ethical Considerations:

All participants will be given an information sheet and have the opportunity to have any questions addressed by the research team. All participants will be required to complete a consent form. If under 16 years, parents will be asked to complete a consent form on behalf of their child. All data collected will be anonymised and stored safely. Data will only be accessible to the research team. Participants will be informed they have the right to withdraw from the study at any point and this will not affect future access to the services provided. Participant who chose to withdraw from the study will have the option for all of their research data to be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* A child or young person with a working or full diagnosis of an Autism spectrum condition (ASC). Parents/carers will be asked to provide proof in the form of a letter that their child has an ASC.
* The child with an ASC must be between the ages of 8-12 years.
* All participants must confirm they are physically fit to participate in this research as some activities involve moderate to vigorous physical activity.
* All children with an ASC who are receiving alternative support are required to declare this prior to participation and specify the type of support received.

Exclusion Criteria:

* Children/young people without a full or working ASC diagnosis
* Children with a full or working diagnosis of ASC not between the ages of 8-12 years
* People who are not deemed physically fit to participate in the activity programme by their own self-assessment.
* Current or recent participation in another clinical trial/study/scientific experiment

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Change in Social Skills Improvement System Rating Scales - Parent (Social Skills Improvement System; Gresham & Elliott (2007). | 14 weeks
  The Social Skills Improvement System (SSIS) evaluates social skills and problem behaviours. Parents/guardians report on the frequency their children exhibit social skills and problem behaviours on a 4-point scale with responses including; 0 'never' , 1 'seldom', 2 'often', and 3 'almost always'. Social skills are evaluated in the following domains: communication, cooperation, assertion, responsibility, empathy, engagement, and self-control. Problem behaviours assessed include: externalizing, bullying, hyperactivity/inattention, internalising, and "autism spectrum". For the social skills domain higher scores indicate better outcomes. For the problem behaviours domain, higher scores indicate poorer outcomes.
Change in Social Skills Improvement System Rating Scales - Child (Social Skills Improvement System; Gresham & Elliott (2007). | 14 weeks
  The Social Skills Improvement System (SSIS) evaluates social skills and problem behaviours. Young people (8-12) indicate if a variety of different statements about problem behaviours or social skills are true of them on a 4-point scale: not true (minimum value), a little true, a lot true, and very true (maximum value). Social skills are evaluated in the following domains: communication, cooperation, assertion, responsibility, empathy, engagement, and self-control. Problem behaviours assessed include: externalizing, bullying, hyperactivity/inattention, internalising, and "autism spectrum". For the social skills domain higher scores indicate better outcomes. For the problem behaviours domain, higher scores indicate poorer outcomes.

SECONDARY OUTCOMES:
Social Connectedness Scale Revised (SCS-R; Lee, Draper & Lee 2001) | 14 weeks
  Social Connectedness is considered is an attribute of the self, reflecting interpersonal thoughts and closeness to the social world. The scale is comprised of 10 negatively worked and 10 positively worded items such as "I feel comfortable in the presence of strangers" and "I feel myself as an outsider". Participants rate the degree to which they agree or disagree on a scale from 1-6 (1= strongly disagree, 6 strongly agree).
Self Image Profile (SIP; Butler) | 14 weeks
  This SIP invites respondents to give two ratings of how they consider themselves to be; and how they would like to be across 25 items. Participants rate each item from 0 (Not At All) to 6 (Very Much). The SIP comprises 12 items of a positive nature i.e. 'Intelligent' and 12 of a negative tone 'mess about'. Once completed a self image score (summation of the first rating) and self esteem score (operationally defined as the discrepancy between the two ratings) can be obtained.
The Short Warwick-Edinburgh Mental Wellbeing Scales (SWEMWBS; Stewart-Brown et al., 2009) | 14 weeks
  The Short version of the Warwick-Edinburgh Mental Wellbeing Scales measures positive aspects of mental health in the prior 2 weeks such as "I've been feeling useful" or "I've been feeling relaxed". The scale comprises 7 positively phrased items responded on a 5-point Likert-type scale from 1 'None of the time' to 5 'All of the time'. Higher scores on this measure indicate a better outcome.
Goal Based Outcomes (GBOs) | 14 weeks
  Parents will be asked to state 3 goals that they wish to achieve from participating in the 10-week programme. Prior to the start of the intervention, parents will be asked to rate where they feel they are now in relation to achieving a specified goal on a scale of 0-10, 0 being 'goal not at all met' and 10 being 'goal reached'. At the end of the intervention, parents will be asked to again rate where they feel they are now in relation to achieving a specified goal on the same rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: James Smolinski, Principal Investigator — Midlands Psychology CIC
Locations (1):
- The Hayes, Stafford, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Butler R.J. (2001) The self-image profile for children (SIP-C) and adolescents (SIP-A). Manual. London, The Psychological Corporation
- [Background] Eccles, J. S., & Barber, B. L. (1999). Student council, volunteering, basketball, or marching band what kind of extracurricular involvement matters? Journal of adolescent research, 14(1), 10-43.
- [Background] Hastings RP, Kovshoff H, Ward NJ, degli Espinosa F, Brown T, Remington B. Systems analysis of stress and positive perceptions in mothers and fathers of pre-school children with autism. J Autism Dev Disord. 2005 Oct;35(5):635-44. doi: 10.1007/s10803-005-0007-8. PMID 16177837
- [Background] Kohl HW 3rd, Hobbs KE. Development of physical activity behaviors among children and adolescents. Pediatrics. 1998 Mar;101(3 Pt 2):549-54. PMID 12224661
- [Background] Lang, R., Koegel, L. K., Ashbaugh, K. et al. (2010). Physical exercise and individuals with autism spectrum disorders: A systematic review. Research in Autism Spectrum Disorders, 4(4), 565-576.
- [Background] Lee, R. M., Draper, M., & Lee, S. (2001). Social connectedness, dysfunctional interpersonal behaviors, and psychological distress: Testing a mediator model. Journal of counseling psychology, 48(3), 310.
- [Background] Neff, K. D., & Faso, D. J. (2015). Self-compassion and well-being in parents of children with autism. Mindfulness, 6(4), 938-947.
- [Background] Memari, A. H., Kordi, R., Ziaee, V. (2012). Weight status in Iranian children with autism spectrum disorders: Investigation of underweight, overweight and obesity. Research in Autism Spectrum Disorders, 6(1), 234-239.
- [Background] Public Health England (2016). Health matters: getting every adult active every day. [online] Available at: https://www.gov.uk/government/publications/health-matters-getting-every-adult-active-every-day/health-matters-getting-every-adult-active-every-day [Accessed 20 Aug. 2019].
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398
- [Background] Trost SG, Kerr LM, Ward DS, Pate RR. Physical activity and determinants of physical activity in obese and non-obese children. Int J Obes Relat Metab Disord. 2001 Jun;25(6):822-9. doi: 10.1038/sj.ijo.0801621. PMID 11439296